CLINICAL TRIAL: NCT00259688
Title: Sleep Disordered Breathing and Preeclampsia
Brief Title: Prevalence Study of Sleep Apnea in Women With Preeclampsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: John Reid - Assistant Professor, University of Saskatchewan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BIO-REB 05-110
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Sleep Apnea; CPAP
MeSH Terms: conditions — Pre-Eclampsia; Sleep Apnea Syndromes

ARMS (3):
- 1 (No Intervention): Women with gestational hypertension
- 2 (No Intervention): Women with uncomplicated pregnancies
  Interventions: Device: CPAP therapy for subjects diagnosed with sleep apnea
- 3 (No Intervention): Re-test of women one to two years post-partum.

INTERVENTIONS:
Device: CPAP therapy for subjects diagnosed with sleep apnea — CPAP therapy is being offered to women who are diagnosed on Polysomnogram with sleep apnea. However, this is not an intervention study and treatment is not part of the study protocol.
  Arms: 2

SUMMARY:
Hypothesis: The prevalence of sleep apnea is greater in pregnant women with preeclampsia than in pregnant women without preeclampsia.The presence of sleep apnea will be associated with poor blood pressure control, worsening blood pressure during sleep and evidence of fetal distress. The usual treatment for sleep apnea is to have the patient breathe pressurized air through a mask. This is called continuous positive airway pressure (CPAP). In preeclamptic women with sleep apnea, use of CPAP will result in improved blood pressure control and reduced fetal distress.

DETAILED DESCRIPTION:
Sleep apnea is common in the adult population. In middle aged men, the presence of sleep apnea has been correlated with hypertension, cardiovascular disease and mood disorders. Sleep apnea is not as well studied in women and even less is known about sleep apnea in pregnant women. However, preliminary evidence suggests that the incidence is quite high, particularly in women with severe preeclampsia. We propose to perform sleep studies on 30 women with preeclampsia and 30 healthy pregnant controls. In addition to the usual sleep study monitoring, we will also measure beat-to-beat blood pressure through non-invasive monitoring and we will do continuous electronic fetal monitoring. Women found to have sleep apnea will have a repeat study in which CPAP therapy is applied, and be provided CPAP therapy for nightly use at home.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women >18 years of age

Exclusion Criteria:

* significant medical conditions that would be expected to affect maternal- fetal outcomes
* need for admission to hospital, so that it transfer to the sleep would compromise maternal-fetal safety

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of sleep apnea in preeclampsia and pregnancy. | Time of delivery for each woman

SECONDARY OUTCOMES:
For those subjects diagnoses with sleep apnea: Improvement in blood pressure and electronic fetal monitoring during with use of CPAP. | Time of delivery for each woman

CONTACTS AND LOCATIONS:
Overall Officials: John K Reid, MD, BSc, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital Sleep Disorders Centre, Saskatoon, Saskatchewan, Canada